## A Randomized Pilot Trial of Dilute Povidone-iodine Irrigation vs No Irrigation for Children with Acute, Perforated Appendicitis

NCT02664220

Version Date: 08/29/2016

# A Randomized Pilot Trial of Dilute Povidone-iodine Irrigation vs No Irrigation for Children with Acute, Perforated Appendicitis

| Site(s) involved and PI name(s) for corresponding site: |
|---|
| University of Texas Health Sciences Center at Houston (Children's Memorial Hermann |
| Hospital): KuoJen Tsao, MD |

#### **Protocol**

Statement of Compliance

Signature Page

List of Abbreviations

Abstract

| 1 | Key l | Roles |
|---|---|---|
| 2 | Back | ground Information and Scientific Rationale |
| | 2.1 | Background Information |
| | 2.2 | Scientific Rationale |
| | 2.3 | Potential Risks and Benefits |
| | | 2.3.1 Potential Risks |
| | | 2.3.2 Known Potential Benefits |
| 3 | Objec | ctives |
| 4 | • | / Design |
| 5 | Study Population | |
| | 5.1 | Selection of the Study Population |
| | 5.2 | Inclusion/Exclusion Criteria |
| 6 Study Procedures/Evalations | | |
| | 6.1 | Study Procedures |
| 7 | Statis | tical Considerations |
| | 7.1 | Study Outcome Measures |
| | 7.2 | Sample Size Considerations |
| | 7.3 | Baysian Prior Probability |
| | 7.4 | Participant Enrollment and Follow-Up |
| | 7.5 | A Priori Practice Algorithm |
| | 7.6 | Analysis Plan |
| | 7.7 | Interim Analysis |
| | 7.8 | Data Safety and Monitoring Board (DSMB) |
| 8 | Subje | ect Confidentiality |
| 9 | _ | med Consent Process |
| 10 | Publi | cation Plans |
| 11 | | rences, Costs, and Funding |
| 12 | Liters | ature References |

#### STATEMENT OF COMPLIANCE

This study will be conducted according to US and international standards of Good Clinical Practice (45 CFR Part 46, 21 CFR Part 50, 21 CFR Part 56, 21 CFR Part 312, and International Conference on Harmonisation guidelines), applicable government regulations, and institutional research policies and procedures.

## **Signature Page**

| KuoJen Tsao, MD |
|------------------------|
| Principle Investigator |

#### **List of Abbreviations**

IAA Intra-abdominal abscess

CMHH Children's Memorial Hermann Hospital

PVI Povidone-iodine (aka. Betadine®)

CT Computed tomography

#### **Significance**

Postoperative intra-abdominal abscesses are common occurrences after perforated appendicitis in pediatric patients despite utilization of evidence-based practices. Povidone-iodine is a commonly used antiseptic in surgical procedures and has been shown to be effective in reducing postoperative abscesses in adults with perforated appendicitis. This trial will be the first to rigorously test the efficacy of povidone-iodine irrigation in children and to verify its safety profile in this patient population.

### 1.0 Key Roles

KuoJen Tsao, MD: As the Principle Investigator, Dr. Tsao will be responsible for the overall study from the surgical and medication administration perspective, compliance with regulations and ethical standards, patient safety, accuracy of the study results and reporting.

#### 2.0 Background Information and Scientific Rationale

#### 2.1 Background

Acute appendicitis is the most common gastrointestinal-related disease requiring surgery in children. Nearly 25% of all children with perforated appendicitis develop postoperative surgical site infections, specifically intra-abdominal abscesses (IAA), which is likely due to the intra-abdominal sepsis that occurs with the perforated viscus [1,2]. These IAA lead to increased patient discomfort, extended hospital stays, and increased emergency room visits and readmissions [3]. In line with other children's hospitals in the country, Children's Memorial Hermann Hospital (CMHH) has implemented evidence-based practices such as early and culture-directed antibiotic coverage, early operation, and protocol-driven postoperative care [1,2]. Specifically for patients with perforated appendicitis, over the course of four years, our dedicated team of pediatric surgeons has reviewed patient outcomes on an iterative basis, leading to targeted intraoperative and postoperative interventions such as transperitoneal drain placement and customized home antibiotic regimens in an attempt to decrease postoperative IAA. Despite all these efforts, the IAA rate has remained unchanged.

In a 2004 survey of North American pediatric surgeons, over 90% responded that they use intraabdominal irrigation for patients with advanced appendicitis [4]. However, although its use is
widespread, intraoperative irrigation has not been widely studied. There is strong evidence of no
difference in IAA rate when no irrigation is compared to normal saline irrigation for children
with perforated appendicitis [5], and there is even some evidence that suggests that NS irrigation
may actually increase the rate of postoperative IAA [6]. Another irrigation solution that is widely
available and commonly used in the operating room is povidone-iodine (PVI). PVI is an
antiseptic solution consisting of polyvinylpyrrolidone with water, iodide, and 1% available
iodine. It has bactericidal ability against a large array of pathogens, including those pathogens
which commonly cause postoperative IAA in children with perforated appendicitis [7,8]. Just a
few examples of how PVI is used for surgery include: skin and mucosal preoperative
preparation, intestinal intraluminal irrigation prior to division and anastomosis, mediastinal
washout following sternal wound infections, and refractory chylothorax in newborns [9–11].



Although PVI is commonly used in pediatric operations, its use as an intra-abdominal irrigant for perforated appendicitis has not been rigorously studied.

A recent meta-analysis demonstrated that intraoperative irrigation with PVI in abdominal, gynecologic, and spinal surgeries significantly decreased postoperative abscesses compared to normal saline irrigation or no irrigation at all (pooled relative risk 0.13, 95%CI 0.05-0.37, p<0.001) [12]. However, of the trials included in this particular analysis, only two of the four focused on treating intra-abdominal sepsis and neither of the studies indicated the number or age of pediatric patients who were enrolled [13,14]. A recent survey of European general adult surgeons found that nearly 40% of them commonly use PVI irrigation for contaminated or dirty abdominal surgeries such as perforated appendicitis [15]. Despite the existing data supporting the efficacy of PVI to reduce IAA and its common use in dirty abdominal surgeries, there have been no recent, high-quality trials demonstrating its effectiveness in reducing IAA after perforated appendicitis in children.

#### 2.2 Scientific Rationale

**Hypothesis:** Among pediatric patients presenting to CMHH with perforated appendicitis, intraabdominal irrigation with PVI versus no irrigation will decrease the rate of 30-day postoperative IAA.

**Specific Aim 1:** To conduct a pilot randomized controlled trial to compare the efficacy of PVI irrigation to no irrigation for decreasing postoperative IAA in children with perforated appendicitis

**Specific Aim 2:** To verify the safety profile of dilute PVI for intra-abdominal irrigation **Specific Aim 3:** To determine the effect of PVI irrigation vs no irrigation on hospital length of stay, readmissions, and cost

#### 2.3 Potential Risks and Benefits

PVI is commonly used in the surgical treatment of adults with dirty abdominal surgeries such as perforated appendicitis [15]. PVI could cause an allergic reaction or iodine toxicity; however, this is exceptionally rare, especially at dilute concentrations [16]. Potential benefits include a reduction in postoperative IAA, decreased length of stay, and fewer readmissions. The



knowledge obtained from this study could help to improve patient outcomes following acute, perforated appendicitis as well as provide preliminary data for a larger, pragmatic trial.

There is a possibility of breach of confidentiality. However, all data collected will be put into a password protected database with will be kept on a pasword-protected secure server with access limited to study personnel assocaited with the study.

3.0 Objectives

To determine the effect of PVI irrigation versus no irrigation on the rate of IAA at 30-days postoperative following appendectomy for acute, perforated appendicitis

4.0 Study Design

This will be a single-center, pilot RCT carried out by the Pediatric Surgery Department at UT Houston – CMHH. All UT Houston pediatric surgery attendings will participate. Patients will be randomized to PVI irrigation or no irrigation.

5.0 Study Population

5.1 Selection of the Study Population

A team of five pediatric surgery research coordinators will coordinate the enrollment, consent, and assent processes. The research coordinator team will be available 24/7 to the pediatric surgery service via a dedicated pager. Residents and attendings on the pediatric surgery service will page the research coordinators upon diagnosing a patient with suspected appendicitis. All patients undergoing appendectomy for acute appendicitis will be eligible for the trial. After enrollment, only patients who are diagnosed intraoperatively with perforated appendicitis will be randomized.

5.2 Inclusion/Exclusion Criteria

*Inclusion criteria:* Patients aged 2-17 years old who undergo an appendectomy for acute, perforated appendicitis at CMHH. Diagnosis of perforated appendicitis is made intraoperatively

IRB NUMBER: HSC-MS-15-1000
UTHealth
The University of Texas

by the surgeon and is defined as the visualization of a gross defect in the appendiceal wall or the

presence of intraperitoneal stool or a fecalith at the time of operation.

Exclusion criteria: 1) patients presenting with simple or gangrenous appendicitis, 2) patients

with a history of iodine sensitivity, thyroid disease or renal disease, 3) patients undergoing

interval or incidental appendectomy, and 4) pregnancy.

We do not anticipate pregnancy in our study population. Pregnant subjects and their fetuses may

be placed at undue risk for the purposes of the study. Therefore, pregnant patients will be

excluded from participating in the study.

Withdrawal: Prior to or after providing informed consent, patients may withdraw from the study

at any point pre- or postoperatively by informing any of the care providers during the patient's

hospital stay.

**6.0 Study Procedures/Evaluations** 

**6.1 Study Procedures** 

Randomization and allocation:

Enrollment will occur prior to the operation either in the emergency room, on the ward, or in the

preoperative holding area. The randomization schema will be variable block randomization, and

sequentially numbered, opaque, sealed envelopes will be used to blind allocation. Following

consent, the sealed, opaque envelope will be attached to the patient's chart which accompanies

the patient into the operating room. Only if the patient is found intraoperatively to have

perforated appendicitis will the envelope be opened by the circulating nurse and the patient

assigned to the control or intervention group. If a patient is determined to have simple or

gangrenous appendicitis, the sealed envelope will remain unopened, and a research coordinator

will retrieve it for re-use.

Standard Preoperative, Operative, and Postoperative Protocols

UTHeath IF
The University of Texas
Health Science Center at Houston

IRB NUMBER: HSC-MS-15-1000 Health IRB APPROVAL DATE: 08/29/2016 Upon patient admission to the hospital, the patient will be started on the preoperative appendicitis protocol that has been in place at CMHH since 2011. Briefly, this protocol entails immediate initiation of intravenous piperacillin-tazobactam or metronidazole/gentamicin for patients allergic to penicillin. The intravenous antibiotics are continued throughout the inpatient admission. Additionally, patients are fluid resuscitated and analgesia is provided.

A laparoscopic approach will be attempted for all patients; however, conversion from laparoscopy to an open technique will not result in exclusion from the trial. After carefully examining the peritoneal cavity and upon identifying the appendix, the surgeon will declare whether or not the patient has a perforated appendicitis (as defined previously). At that point, the circulating nurse will open the sealed envelope and group assignment will occur. Subsequently, once the surgeon has removed the appendix from the abdomen and ensured hemostasis, the surgeon will proceed to use the battery-powered, suction-irrigator device to irrigate primarily the right upper, right lower, and pelvic regions as these are the predominant locations for postoperative IAA formation [5]. If the patient is assigned to the intervention group, the nurse will create the dilute PVI irrigation by first removing 100ml of saline from a 1000ml bag and replacing it with 100ml of stock, 10% PVI (readily available in the operating room), thereby creating an irrigation solution with 1% PVI. Dilution of the PVI will occur while the surgeon completes the operation (removes the appendix). Once the appendix has been removed and hemostasis ensured, the surgeon will perform the irrigation with 10cc/kg (minimum 100ml and maximum 1000ml) of dilute PVI. The dose of PVI (10cc/kg) is based on previous studies [13,14] as well as consensus from our pediatric surgery team and is felt to be a conservative dose [14]. After completing the irrigation, the surgeon will suction out all intra-abdominal fluid into a suction canister and the amount will be recorded. Patients allocated to the control group will not undergo intra-abdominal irrigation.

All postoperative care will follow the standardized perforated appendicitis care pathway which includes continued intravenous antibiotics until they are discharged from the hospital. Standard discharge criteria for perforated appendicitis patients will comprise the following parameters: oral/axillary temperature < 100°F (oral) x 24hr, tolerating regular diet, pain relief with oral analgesics, ambulating with minimal assistance as age appropriate, normal white blood cell count

without bandemia. Those patients who do not meet discharge criteria within seven days will undergo a computed tomography (CT). Patients diagnosed with an IAA on CT scan will receive an interventional radiology consultation and will undergo percutaneous drainage when deemed feasible by the interventional radiologist.

The same discharge criteria will apply for all patients. All patients will be scheduled for follow-up with a pediatric surgeon within one week of discharge. Those patients who are not able to attend the follow up appointment will be called and rescheduled. In the clinic, a post-appendectomy form (Appendix A) will be filled out by a pediatric surgeon who will document physical exam findings as well as any additional postoperative complications or visits to an emergency room (ER) or other healthcare facility as reported by the patient/parents. All patients will be called between 30-32 days postoperatively (in case postoperative day 30 falls on the weekend), and a form will be filled out that details any further complications or healthcare facility visits.

Postoperative Laboratory Testing & 6- and 12-month Follow Up

To verify the safety profile of PVI irrigation, at the time of intraoperative diagnosis of perforated appendicitis, the anesthesia provider will send a blood sample to the lab to measure baseline glucose, TSH, and T4 levels in 10 patients. Two additional samples will be sent at 24 hours and as needed at 72 hours postoperatively by the floor nurse. Pediatric endocrinology will follow these first 10 patients during their admissions and will provide therapeutic guidance in the unlikely event that symptomatic hypothyroidism occurs. Six and 12-month follow up with patients (via chart review and phone call) will take place to determine if any small bowel obstructions occur due to abdominal adhesions. Although rare, abdominal adhesions are a known entity after appendectomy and theoretically may be exacerbated by either normal saline or PVI irrigation.

#### 7.0 Statistical Consideration

Providing both frequentist and Bayesian approaches has been shown to provide complementary interpretations [17]. Furthermore, while a frequentist analysis may result in a "negative" study, posterior probabilities based on a Bayesian approach may still be sufficient for clinicians to



implement an intervention despite an insignificant p-value or to recruit additional centers to participate in an ongoing study. There are several more reasons why performing a Bayesian analysis alongside a frequentist analysis may be beneficial, many of which are listed in a study by Wijeysundera and colleagues [17]. Therefore, our study will include both frequentist and Bayesian analyses.

#### 7.1 Study Outcome Measures

The primary outcome will be 30-day postoperative IAA rate. An IAA will be defined as an image-confirmed (ultrasound or CT) fluid collection deemed to be an IAA by a pediatric radiologist at CMHH. The imaging studies will be obtained for patients who undergo postoperative imaging at outside facilities and will be read by CMHH pediatric radiologists. The radiologists will remain blinded to the patient's intervention. Patients who are determined to have an IAA will be referred to interventional radiology for percutaneous drainage and will be restarted on intravenous antibiotics based on organism susceptibilities.

Secondary outcomes will include total hospital length of stay within 30 postoperative days and rates of readmissions and ER visits within 30 postoperative days. Total hospital length of stay will be the aggregate of all days in the hospital including any appendicitis-related readmissions within 30 postoperative days. Thirty-day ER visits and readmissions will also be determined through chart review, clinical encounters, and phone calls. Other adverse events that will be recorded will include abnormal thyroid function tests requiring endocrinology intervention immediately postoperatively and small bowel obstructions within one year after surgery.

A small outcomes adjudication committee will review a random sample of patient charts to verify the reported findings. Members of the committee will have no vested interest in the outcomes of the proposed study and will be blinded to treatment allocation.

The patient list will be generated when the pediatric surgery team informs the research coordinator that a patient with suspected appendicitis is being consented for an appendectomy. The patient MRN will be converted to a unique patient ID using a linking log that is accessible to the study coordinators. Electronic records from Children's Memorial Hermann Hospital and UT



professional building pediatric surgery clinic will be accessed. The data will be collected by the principle investigator and those listed in the IRB application. No patient identifiers will be collected. Data points to be abstracted from the electronic medical record or requested from the Memorial Hermann Hospital system will include:

- 1. Age
- 2. Race
- 3. Gender
- 4. Height
- 5. Weight
- 6. Admission date(s)
- 7. Admission time(s)
- 8. Admission location(s)
- 9. Discharge date(s)
- 10. Discharge time(s)
- 11. OR date(s)
- 12. Postoperative diagnosis
- 13. Operative procedures
- 14. Operative reports
- 15. Pathologic diagnosis
- 16. Laboratory results
- 17. Imaging type(s)
- 18. Imaging dates(s)
- 19. Imaging location(s)
- 20. Imaging results
- 21. Dates and causes of any readmissions
- 22. Medications administered, including antibiotics
- 23. Administration dates of medications
- 24. Side effects related to antibiotic administration
- 25. Dates of diet advancement
- 26. Date(s) of surgical site infections



27. Hospital costs (to be requested from the Memorial Hermann Hospital system)

a. Direct and indirect costs associated with hospital stay

7.2 Sample Size Considerations

Using a frequentist approach, to demonstrate a clinically important decrease in IAA from 24% to 16% with 80% power and a two-tailed significance level of 0.05, a sample size of 784 patients (392 patients per group) would be required. Based on current practice (approximately 100 appendectomies are performed annually for perforated appendicitis) and an estimated consent

rate of 50%, study enrollment would take approximately 15 years.

In anticipation of using a Bayesian approach, the CMHH pediatric surgeons have come to consensus that they would change the way they practice if a Bayesian analysis could determine with 75% confidence whether or not PVI is beneficial. Based on Monte-Carlo simulations using the prior probabilities described below, our pediatric surgeons are confident that a 2-year, pilot

trial will provide sufficient power to guide future efforts (Appendix B).

7.3 Bayesian Prior Probabilities

A Bayesian prior represents the probability distribution that summarizes the beliefs about the treatment benefit prior to seeing study results. The prior is determined by taking into account existing evidence, expert knowledge and option, and defining clinically important outcomes. After thorough review of the current literature concerning intra-abdominal irrigation for perforated appendicitis (which are referenced in the Introduction) and discussion, the CMHH pediatric surgeons feel the following Bayesian priors are appropriate for analyzing the benefit of PVI in this trial (RR=relative risk, CI=confidence interval):

Neutral: RR 1 (95%CI 0.5-1.6) Optimistic: RR 0.67 (95%CI 0.3-1.2)

24% IAA (95%CI 13-37%) 16% IAA (95%CI 9-34%)

To determine the prior probability of treatment benefit for the control group (no irrigation), we will use three years of prospectively collected data from CMHH of patients who underwent the current protocol which is to not perform irrigation (n=325). Further strengthening this prior

17



probability is the fact that similar results have been published by similar programs across the country [1,2]. The following prior will be used when analyzing the benefit of no irrigation (control group) during the trial: 24% IAA (95%CI 20-29%)

#### 7.4 Participant Enrollment and Follow-Up

A multidisciplinary, post-appendectomy surveillance program developed by the Infection Control and Pediatric Surgery departments has been in place since 2011 and is tasked with prospective surveillance of all appendicitis patients. Through the joint efforts of both departments, all appendicitis patients are closely followed during the 30 days after discharge through electronic medical record review, wound culture review, and all SSI reporting among the Memorial Hermann Hospital affiliates (11 hospitals in the Houston metropolitan area). Each documented SSI is jointly reviewed by members of both departments during a monthly meeting.

#### 7.5 A Priori Practice Algorithm

The CMHH pediatric surgeons have devised an *a priori* algorithm to guide their next steps in clinical practice based on the study results at the end of two years. The algorithm uses an optimistic prior probability of treatment success and takes into account the results of the Monte-Carlo simulations previously performed (Appendix B).



7.5 Analysis Plan

Demographics and baseline characteristics of each group will be clearly displayed in a table.

Primary and secondary outcomes will be determined and compared for each group, including

effect sizes and 95% CI. For binary outcomes, absolute and relative effect sizes will be

determined. Bayesian probability models will also be performed to determine the likelihood and

degree of treatment benefit. Chi-square, Fisher's exact, Student's t-test or Mann-Whitney U tests

will be performed for categorical and continuous variables, respectively. Generalized linear

models will be utilized to look at predictors of IAA, ER visits, readmissions, and LOS. The data

will be analyzed based on their distribution.

A CONSORT flow diagram will be provided to clearly demonstrate the number of participants

who were randomized, received the intended treatment, and were analyzed for the primary and

secondary outcomes. The reasons for losses to each group will be documented; intention-to-treat

(primary) and per-protocol (secondary) analyses will be performed.

Limitations

(1) Subjectivity of the primary outcome. An outcome such as IAA may be subjective due to

variable definitions or interpretations. However, we utilized a standardized definition that is

utilized, endorsed, and has been validated by other pediatric surgeons [18]. In addition, trained

clinicians blinded to the allocation will make the assessments.

(2) Failure to blind the treating clinicians. Clinicians making treatment decisions may not be

blinded to the intervention if they were present during the operation. However, postoperative

protocols are in place to help minimize differential treatment based on treatment allocation.

Additionally, the patients, radiologists, and data analysts will be blinded. Research coordinators

will keep a separate spreadsheet to keep track of group assignment.

(3) Generalizability. This study will be performed on pediatric patients at a tertiary care

academic center. The applicability of these results to other clinical settings may be limited. If this

UTHealth
The University of Texas

study demonstrates safety and efficacy, other institutions will be recruited for a larger, multicenter trial.

7.7 Interim Analysis

Six months after the first patient is enrolled, an interim analysis will be conducted by an independent Data & Safety Monitoring Board to ensure there are no increased harms of PVI and that ongoing study participation is not futile.

7.8 Data Safety and Monitoring Board (DSMB)

The DSMB will be composed of a general surgeon, pediatric endocrinologist, infectious disease physician, statistician, and an academic surgeon with clinical trial experience.

Harms will entail but not be limited to: abnormal thyroid tests requiring endocrinology intervention or adhesive small bowel obstruction requiring readmission or surgery. There are no other anticipated harms imposed by PVI irrigation; however, any unexpected harms that arise will be included in the interim and final analyses. At the time of the interim analysis, if the probability of increased harms is >75% or the probability that PVI is beneficial is <10%, the study will be stopped and existing data will be reported.

8.0 Subject Confidentiality

Patient data will be entered into a secure, UT-Houston REDCap database [19] by the study coordinators. Only study investigators approved by the Institutional Review Board to participate in the study will have access to the REDCap data. Upon completion of the study, the REDCap database will be permanently deleted.

9.0 Informed Consent Process

Consent will be obtained from each participant prior to surgery after verification that all inclusion and exclusion criteria have been met. Patients will have the consent read to them by one of the coordinators and all questions will be answered. Minors will also be assented for the study. Subjects who speak languages other than English will be commnicated with using an official interpreter via the Hermann translator line. This will allow the research team the

IRB NUMBER: HSC-MS-15-1000
UTHealth IRB APPROVAL DATE: 08/29/2016

opportunity to discuss the consent, answer and questions and discuss the protocol with the assistance of a certified interpreter. All patients willing to be enrolled in the study will receive a signed copy of the consent form.

A Waiver of Consent will be requested for eligible study participants unable to provide assent or parents/guardians who refuse to sign an informed consent for the following reasons:

- Emergent intervention requiring medical sedation, incapacitation, and/or endotracheal intubation (i.e. septic shock, cardiopulmonary resuscitation)
- Auditory, visual, or mental impairment and/or learning disability
- Parent or guardian preference refusal or declination to permit child to provide assent (i.e. extreme fatigue, weakness, lethargy)

#### 10.0 Differences, Costs, and Funding

Currently, each arm of the study (PVI or no irrigation) has been deemed to be safe and is utilized commonly by some surgeons in some settings as the standard of care. The unique portion of the intervention is simply randomizing all of the interventions in a systematic fashion rather than in a arbitrary fashion (current practice).

We do not feel that any of the interventions or follow-ups represent a cost to the patient or healthcare system above current practice.

Currently, we are seeking funding to support this trial. However, without an IRB number and approved IRB, many funding sources are not available. We anticipate seeking funding from intra- and extra-mural grants.

#### **Literature References**

- [1] Blakely ML, Williams R, Dassinger MS, Eubanks JW, Fischer P, Huang EY, et al. Early vs interval appendectomy for children with perforated appendicitis. JAMA Surg 2011;146:660–5.
- [2] St Peter SD, Aguayo P, Fraser JD, Keckler SJ, Sharp SW, Leys CM, et al. Initial laparoscopic appendectomy versus initial nonoperative management and interval



- appendectomy for perforated appendicitis with abscess: a prospective, randomized trial. J Pediatr Surg 2010;45:236–40.
- [3] Newman K, Ponsky T, Kittle K, Dyk L, Throop C, Gieseker K, et al. Appendicitis 2000: variability in practice, outcomes, and resource utilization at thirty pediatric hospitals. J Pediatr Surg 2003;38:372–9; discussion 372–9.
- [4] Muehlstedt SG, Pham TQ, Schmeling DJ. The management of pediatric appendicitis: a survey of North American Pediatric Surgeons. J Pediatr Surg 2004;39:875–9.
- [5] St Peter SD, Adibe OO, Iqbal CW, Fike FB, Sharp SW, Juang D, et al. Irrigation versus suction alone during laparoscopic appendectomy for perforated appendicitis: a prospective randomized trial. Ann Surg 2012;256:581–5.
- [6] Moore C, Smith R, Herbertson R, Toevs C. Does Use of Intraoperative Irrigation with Open or Laparoscopic Appendectomy Reduce Post-Operative Intra-abdominal Abscess? Am Surg 2011;77:78–80.
- [7] Zamora JL, York N. Chemical and Microbiologic Characteristics and Toxicity of Povidone-Iodine Solutions 1956.
- [8] Fallon SC, Hassan SF, Larimer EL, Rodriguez JR, Brandt ML, Wesson DE, et al. Modification of an evidence-based protocol for advanced appendicitis in children. J Surg Res 2013;185:273–7.
- [9] Parker M, EC A, MWN N, CH D, JC B. Povidone-iodine colorectal carcinoma. Ann R Coll Surg Engl 1985;67:1–2.
- [10] Kovacikova L, Kunovsky P, Skrak P, Hraska V, Kostalova L, Tomeckova E. Thyroid hormone metabolism in pediatric cardiac patients treated by continuous povidone-iodine irrigation for deep sternal wound infection. Eur J Cardiothorac Surg 2002;21:1037–41.
- [11] Scottoni F, Fusaro F, Conforti A, Morini F, Bagolan P. Pleurodesis with povidone–iodine for refractory chylothorax in newborns: Personal experience and literature review. J Pediatr Surg 2015.
- [12] Fournel I, Tiv M, Soulias M, Hua C, Astruc K, Glele LSA. Meta-analysis of intraoperative povidone-iodine application to prevent surgical-site infection. Br J Surg 2010;97:1603–13.
- [13] Sindelar WF MR. Intraperitoneal Irrigation with Povidone-Iodine Solution for the Prevention of Intra-abdominal Abscesses in the Bacterially Contaminated Abdomen. Surg

- Gynecol Obstet 1979;148:409-11.
- [14] Sindelar WF, Brower ST, Merkel AB, Takesuet EI. Randomised trial of intraperitoneal irrigation with low molecular weight povidone-iodine solution to reduce intra-abdominal infectious complications. J Hosp Infect 1985;6:103–14.
- [15] Whiteside OJH, Tytherleigh MG, Thrush S, Farouk R, Galland RB. Intra-operative peritoneal lavage--who does it and why? Ann R Coll Surg Engl 2005;87:255–8.
- [16] Lachapelle JM. A comparison of the irritant and allergenic properties of antiseptics. Eur J Dermatology 2014;24:3–9.
- [17] Wijeysundera DN, Austin PC, Hux JE, Beattie WS, Laupacis A. Bayesian statistical inference enhances the interpretation of contemporary randomized controlled trials. J Clin Epidemiol 2009;62:13–21.e5.
- [18] St Peter SD, Sharp SW, Holcomb GW, Ostlie DJ. An evidence-based definition for perforated appendicitis derived from a prospective randomized trial. J Pediatr Surg 2008;43:2242–5.
- [19] Harris P a, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform 2009;42:377–81.

## Appendix A: Pediatric Appendicitis, Standardized Clinical Follow-up Form

| | 14 day | ion Form □ 30 day | |
|---|---|---|---|
| Date of Clinic visit: | 06/04/19 | | |
| Date of Discharge: | 05/22/14 | | |
| Was there an in-patient | post-operative in | ntra-abdomina | al infection DYES AND |
| Wound evaluations: | (check all that apply | ,) | |
| Site | No infection | <u>Cellulitis</u> | Dire Calant - L |
| Right lower quadrant | NO IIII CCIOII | Centinus | Pus Stitch abscess |
| Umbilical port | . 0 | | 7 |
| Suprapubic | | | |
| eft lower quadrant port | Or . | | |
| Other | | | 0 0 |
| reatments: (check all th | nat apply) | | |
| None | | | |
| □ Opened wor | ind (culture all open | wounds, not skin. | |
| □ Oral antibiot | ics | | |
| 1° line (with | out history of MF | RSA) | |
| - Cephalexin<br>Dispens | (Keflex) 25 mg/kg/dos<br>ed: 100mg/ml 125mg | e q 12 hours (ma | x dose 4 g/day) for 10 days<br>r 1 gm, Caps 250 or 500 mg |
| 2nd line (wit | h history of MRS/ | 4) | |
| - Clindamycin | 10 mg/kg/dose q 8 h | ours (max dose 1 | .8g/day) for 10 days |
| □ Admitted fro | ed: 75 mg/5ml, Caps 7 | 5mg, 150 mg, 30 | Omg |
| - Admitted II c | HI CHING | | |
| omments: (Examples: Wa | s infection treated by | pediatrician? Wa | s admitted to another hospital?) |

#### **Appendix B: Monte-Carlo simulations**

#### Scenario 1:

- Sample size: n=100 (50/group)
- True IAA rate (no irrigation): 24% (20-29%)
- True IAA rate (PVI): 16% (95%CI 9-34%), RR 0.67 (95%CI: 0.3-1.2)
- 75% posterior probability the RR<1
- Optimistic prior: RR 0.67 (95% CI: 0.3-1.2)
  - $\rightarrow$  89% power

#### Scenario 2:

- Sample size: n=200 (100/group)
- True IAA rate (no irrigation): 24% (20-29%)
- True IAA rate (PVI): 16% (95%CI 9-34%), RR 0.67 (95%CI: 0.3-1.2)
- 75% posterior probability the RR<1
- Optimistic prior: RR 0.67 (95% CI: 0.3-1.2)
  - $\rightarrow$  94% power

#### Scenario 3:

- Sample size: n=100 (50/group)
- True IAA rate (no irrigation): 24% (20-29%)
- True IAA rate (PVI): 16% (95%CI 9-34%), RR 0.67 (95%CI: 0.3-1.2)
- 75% posterior probability the RR<1
- Neutral prior: RR 1 (95% CI: 0.5-1.6)
  - $\rightarrow$  64% power

